CLINICAL TRIAL: NCT00229840
Title: Advanced MR Imaging Evaluation Of Neurosurgical Candidates With Focal Abnormalities
Brief Title: Evaluation of Functional MRI and DTI (Imaging Techniques) in Children With Epilepsy and Focal Brain Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Healthcare of Atlanta (Other)
Responsible Party: Richard Jones, PhD, Children's Healthcare of Atlanta
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Functional MRI
Record Dates: First submitted 2005-09-13; First posted 2005-09-30 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Epilepsy
Keywords: MRI, fMRI, Epilepsy, Pediatric
MeSH Terms: conditions — Epilepsy | interventions — Diffusion Tensor Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Functional MRI, Diffusion Tensor Imaging

SUMMARY:
This study is being done to look at the relationship between brain structure and brain function in patients with epilepsy or focal brain lesions (abnormal areas) that require surgery. This study will look at an imaging technique called magnetic resonance imaging (MRI) for looking at the brain. Specifically, the study will look at functional MRI, which is an imaging technique that can map brain function by taking pictures of the brain as it performs different tasks such as reading, thinking, or moving a body part and diffusion tensor imaging (DTI), which will look at brain structure. These types of imaging may help us learn more about different areas of the brain and how those areas of the brain are used in children with epilepsy. We plan to study 30 children with epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* children with intractable epilepsy

Exclusion Criteria:

* children requiring sedation for scanning

Ages: 4 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2006-02; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Jones, PhD, Principal Investigator — Emory University/Children's Healthcare of Atlanta
Locations (1):
- Children's Healthcare of Atlanta at Scottish Rite, Atlanta, Georgia, United States